CLINICAL TRIAL: NCT03669614
Title: A Phase 1/2a Randomized, Double-Blind, Two-Part, Dose-Ascending, Multicenter Study of the Safety and PK of AR-501 (Gallium Citrate), Administered Via Inhalation, in Healthy Adult and P. Aeruginosa Infected Cystic Fibrosis Subjects
Brief Title: SAD and MAD of Inhaled AR-501 in Health Adults and P. Aeruginosa Infected Cystic Fibrosis Subjects
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aridis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-501-001
Record Dates: First submitted 2018-08-30; First posted 2018-09-13 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Gallium Citrate; Pseudomonas Aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Intervention Model Description: This study is a dose-escalation, placebo-controlled study where subjects are randomized to receive study drug or placebo.
  SAD and MAD HV Phases: The HV SAD and MAD will each include up to 24 adult subjects in 3 groups (8 per dose group) in each the SAD and MAD phase . All subjects will be randomly assigned in a 3:1 ratio to receive a single administration of active drug (12 HVs) or placebo (4 HVs).
  The CF MAD will evaluate 4 different dose levels in a total of 54 adult CF subjects (10 per dose level). The first 3 subjects (sentinel subjects) in the low, medium and high dose level will be randomly assigned at a 2:1 ratio to receive either AR-501 or placebo, for a total of 9 CF subjects. An expanded cohort will randomize 30 adult subjects at a 2:3:3:2 ratio to three doses of inhaled AR-501 or placebo. Subsequently an 80mg Ga dose (top dose) cohort will randomize subjects at a 2:1 ratio to receive either AR 501 or placebo for a total of 15 subjects , including 6 sentinel subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a standard double-blind randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AR-501 inhaled (Experimental): Four doses (low, medium, high, top) of inhaled AR-501 will be used.
  Interventions: Drug: Inhaled AR-501
- inhaled AR-501 Placebo (Placebo Comparator): Four doses (low, medium, high, top) of inhaled placebo will be used
  Interventions: Drug: Inhaled Placebo

INTERVENTIONS:
Drug: Inhaled AR-501 — single and multiple ascending doses of inhaled AR-501
  Other Names: Inhaled Gallium Citrate
  Arms: AR-501 inhaled
Drug: Inhaled Placebo — single and multiple ascending doses of inhaled placebo
  Other Names: Control (inhaled placebo)
  Arms: inhaled AR-501 Placebo

SUMMARY:
This is a Phase 1/2a randomized, double-blind, two-part, dose-ascending, multicenter study of AR-501 (gallium citrate) solution, administered via inhalation, in healthy adult and P. aeruginosa infected cystic fibrosis (CF) subjects. Phase 1 of the study in HV subjects will consist of a single-ascending-dose (SAD) cohort, followed by the HV multiple-ascending-dose (MAD) cohort. Phase 2a of the study in CF subjects will consist of a MAD study design. The study will evaluate the safety and pharmacokinetic (PK) profile of single and repeat administrations of inhaled AR-501 solution in healthy adults, and the safety, PK and efficacy of repeat administrations of inhaled AR-501 solution in P. aeruginosa infected CF subjects.

DETAILED DESCRIPTION:
Three dose levels (low, medium and high) will be assessed in succession, first in healthy volunteer (HV) subjects, then four ascending doses will be assessed in cystic fibrosis (CF) subjects. The study will be performed in 2 parts: Phase 1 part of the study in HV subjects will consist of a single-ascending-dose (SAD) cohort, followed by the HV multiple-ascending-dose (MAD) cohort. Phase 2a part of the study in CF subjects will consist of a MAD study design.

The HV cohort will include up to 48 subjects. The CF cohort will have 54 subjects. Thus, the total number of subjects is 102.

The Phase 1 HV study will be performed at a Phase 1 Clinical Study Unit and the Phase 2a will be performed at approximately 24 clinical trial sites located in the United States and possibly in Europe, some of which may be part of the Cystic Fibrosis Foundation (CFF)-accredited Therapeutic Development Network (TDN) or the European Cystic Fibrosis Society Clinical Trial Network (ECFS-CTN). Subjects who meet all eligibility criteria, including giving informed consent, will be enrolled and undergo a screening period of 28 days for HV cohorts and 42 days for CF Cohorts.

The HV cohort will include up to 24 adult subjects in 3 dose groups (8 per dose group [Low, Medium and High]) for the SAD phase of the study. In each dose group, subjects will be randomly assigned in a 3:1 ratio to the active drug or placebo, resulting in 6 subjects receiving inhaled AR-501 and 2 receiving inhaled placebo in a double-blind manner. The HV MAD phase of the study will include 24 adult subjects in 3 dose groups (8 per dose group [Low, Medium and High]). In each dose group, subjects will be randomly assigned in a 3:1 ratio to active study drug or placebo, resulting in 6 subjects receiving inhaled AR-501 and 2 receiving inhaled placebo in a double-blind manner. All subjects in HV MAD cohorts will receive once weekly inhaled study drug (either AR-501 or matching placebo) for 4 weeks for a total of 5 doses.

The CF MAD cohort will evaluate 4 different dose levels for a total of 54 adult CF. Of the 54 subjects, 40 will be randomized to receive one of the three ascending doses of AR-501, while 14 will be randomized to receive placebo. All subjects in CF cohorts will receive once weekly inhaled study drug (either AR-501 or matching placebo) for 2 weeks for a total of 3 doses.

The primary purpose of this study is to assess preliminary clinical safety of inhaled AR-501. The true frequency of AEs is unknown, and the sample size cannot be estimated accurately. For unknown AEs, the probabilities of observing at least 1 AE among 36 total healthy adult subjects and 40 adult CF subjects receiving any AR-501 dose are ≥ 80% if the true rate of such events are at least 4.4% and 4.8% respectively.

ELIGIBILITY:
Inclusion Criteria (HV Subjects):

1. Written informed consent given by the subject.
2. At least ≥ 18 years old and < 50 years of age.
3. Healthy with no acute medical condition for ≥ 2 weeks prior to screening and no known chronic medical condition requiring regular medical follow up and care.
4. Body mass index (BMI) between 18 and 30 kg/m2, inclusive.
5. Currently nonsmoking and no history of using nicotine/tobacco-containing products for ≥ 5 years prior to screening.
6. Normal chest X-ray, per opinion of the Investigator.
7. FEV1 ≥ 80% of predicted values.
8. No history or current illicit, pharmaceutical drug or alcohol abuse within ≤ 5 years prior to screening.
9. A female subject must meet one of the following criteria:

   If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first administration of the study medication, during the study, and for at least 90 days after the last dose of the study medication. An acceptable method of contraception includes one of the following:
   * Abstinence from heterosexual intercourse
   * Hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
   * Intrauterine device (with or without hormones), OR
   * Agrees to use a double barrier method (e.g., condom and spermicide) during the study and for at least 90 days after the last dose of the study medication

   If a female of non-childbearing potential, the subject should be surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses), as confirmed by follicle stimulating hormone (FSH) levels.
10. A male subject must agree to use a double barrier method (e.g., condom and spermicide) during the study and for at least 90 days after the last dose of the study medication.

Inclusion Criteria (CF Subjects):

1. Written informed consent given by the subject.
2. At least18 years old
3. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   * Sweat chloride equal to or greater than 60 mmol/liter by quantitative pilocarpine iontophoresis test (QPIT)
   * Two well-characterized, disease-causing mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene.
4. Confirmation of current colonization/infection with P. aeruginosa defined as: a positive sputum or oropharyngeal swab culture at screening.
5. Respiratory symptoms and CF status are stable with no acute exacerbation at the time of randomization.
6. BMI ≥ 18 kg/m2
7. Currently non-smoking and no history of using nicotine/tobacco-containing products or smoking/vaping (inhaled tobacco products or other inhaled substances) for ≥ 1 year prior to screening.
8. FEV1 ≥ 45% of predicted values.
9. Serum creatinine and total bilirubin are both < 1.5 x upper limit of normal (ULN) range (isolated bilirubin > 1.5 x ULN range is acceptable if bilirubin is fractionated and direct bilirubin is < 35%).
10. A female subject must meet one of the following criteria:

    * If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 21 days prior to the first administration of the study medication, during the study, and for at least 28 days after the last dose of the study medication. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
      * Intrauterine device (with or without hormones), OR
      * Agrees to use a double barrier method (e.g., condom and spermicide) during the study and for at least 28 days after the last dose of the study medication
    * If a female of non-childbearing potential, the subject should be surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses), as confirmed by FSH levels.
11. A male subject must agree to use a double barrier method (e.g., condom and spermicide) during the study and for at least 28 days after the last dose of the study medication.
12. Ability to produce an oropharyngeal sample (e.g., Expectorated Sputum or throat swab).

Exclusion Criteria (HV Subjects):

None of the following criteria can be met.

1. Female subjects who are currently pregnant or lactating.
2. Oral temperature above 37.5ºC at the time of screening or prior to randomization.
3. Clinically abnormal renal function, evidenced by serum creatinine > 1.5 mg/dL.
4. Need for using any nephrotoxic agents during the study.
5. Known allergy or hypersensitivity to albuterol.
6. Significantly abnormal liver function:

   1. Total bilirubin >1.5 x upper limit of the normal range (ULN),
   2. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3 x ULN and alkaline phosphatase (ALP) > 2 x ULN
7. Hemoglobin <10 g/dL
8. Abnormal corrected serum calcium concentration prior to enrollment.
9. History or current use of illicit, pharmaceutical drug or alcohol abuse within 5 years prior to screening.
10. Positive urine screen for alcohol, cotinine and/or drugs of abuse at screening and admission.
11. Positive test results for Human Immunodeficiency Virus (HIV)-1/HIV-2 antibodies, Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibody (HCVAb).
12. Inability to comply with any study requirements based on judgement of the Investigator.
13. Any medical, psychological, cognitive, social or legal conditions that would interfere in the ability to give an informed consent and/or participate fully in the study.
14. Participation in another clinical trial involving receipt of an investigative product within 30 days before screening.
15. Any other reason as determined by an Investigator.

Exclusion Criteria (CF Subjects):

None of the following criteria can be met.

1. Female subjects who are currently pregnant or lactating.
2. Oral temperature above 37.5ºC (or temporal temperature above 38.0ºC) at the time of screening or prior to randomization.
3. Serum creatinine > 1.5 mg/dL or known significant kidney disease.
4. Significantly abnormal liver function:

   1. Total bilirubin > 1.5 x ULN range,
   2. ALT and/or AST > 3 x ULN range and ALP > 2 x ULN range.
5. History of medically attended hemoptysis < 1 year (small amount of blood streaking in sputum is acceptable).
6. Pulmonary exacerbations within 3 months prior to randomization (defined as requiring IV antibiotics), in the hospital or at home.
7. Hemoglobin < 10 g/dL.
8. Abnormal corrected serum calcium concentration prior to randomization (normal range is typically 8.5-10.2 mg/dL).
9. Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or re-initiation) in a chronic treatment/prophylaxis regimen for CF or CF-related conditions within 2 weeks prior to randomization.
10. Known allergy or hypersensitivity to albuterol or any component of the study drug or placebo
11. Use of illicit, pharmaceutical drug or alcohol abuse within 6 months prior to screening.
12. Positive urine screen for alcohol, cotinine and/or drugs of abuse at screening (positive results for a subject on Orkambi should have a confirmatory test for cannabinoids performed, e.g., reflex testing, to rule out cross reaction with Orkambi).
13. History of positive test result for human immunodeficiency virus (HIV) HIV-1/HIV-2 antibodies, HBsAg or chronic hepatitis C virus infection.
14. Inability to comply with any study requirements based on judgement of the Investigator.
15. Any medical, psychological, cognitive, social or legal conditions that would interfere in the ability to give an informed consent and/or participate fully in the study.
16. Participation in another clinical trial involving receipt of an investigative product within 30 days before randomization.
17. Suspected or confirmed acute respiratory infection (Examples: bacterial pneumonia, influenza, COVID-19).
18. Any other reason as determined by an Investigator.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Clinical safety profile (adverse events) - Single Ascending Dose | 28 days following dose administration
  Evaluation of adverse events in HV subjects
Clinical safety profile (adverse events) - Multiple Ascending Dose | up to 28 days after last dose administration
  Evaluation of adverse events in HV and CF subjects

SECONDARY OUTCOMES:
Pharmacokinetics (PK) Profile - SAD Cmax | 28 days following dose administration
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: Observed maximum concentration (Cmax)
Pharmacokinetics (PK) Profile - SAD Tmax | 28 days following dose administration
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: time to reach maximum concentration (Tmax)
Pharmacokinetics (PK) Profile - SAD AUC0-inf | 28 days following dose administration
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: area under the time-concentration curve (AUC) from time zero to infinity (AUC0-inf)
Pharmacokinetics (PK) Profile - SAD AUC0-last | 28 days following dose administration
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: area under the time-concentration curve (AUC) from time zero to the last dose (AUC0-last)
Pharmacokinetics (PK) Profile - SAD λz | 28 days following dose administration
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: terminal elimination rate (λz)
Pharmacokinetics (PK) Profile - SAD t½ | 28 days following dose administration
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: half-life (t½)
Pharmacokinetics (PK) Profile - SAD Clp | 28 days following dose administration
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: plasma clearance (Clp)
Pharmacokinetics (PK) Profile - MAD Cmax | up to 28 days after last dose administration
  Pharmacokinetics Characteristics in Multiple Ascending Dose CF Subjects: Observed maximum concentration (Cmax)
Pharmacokinetics (PK) Profile - MAD Tmax | up to 28 days after last dose administration
  Pharmacokinetics Characteristics in Multiple Ascending Dose CF Subjects: time to reach maximum concentration (Tmax)
Pharmacokinetics (PK) Profile - MAD AUC0-inf | up to 28 days after last dose administration
  Pharmacokinetics Characteristics in Multiple Ascending Dose CF Subjects: area under the time-concentration curve (AUC) from time zero to infinity (AUC0-inf)
Pharmacokinetics (PK) Profile - MAD AUC0-last | up to 28 days after last dose administration
  Pharmacokinetics Characteristics in Multiple Ascending Dose CF Subjects: area under the time-concentration curve (AUC) from time zero to the last dose (AUC0-last)
Pharmacokinetics (PK) Profile - MAD λz | up to 28 days after last dose administration
  Pharmacokinetics Characteristics in Multiple Ascending Dose CF Subjects: terminal elimination rate (λz)
Pharmacokinetics (PK) Profile - MAD t½ | up to 28 days after last dose administration
  Pharmacokinetics Characteristics in Multiple Ascending Dose CF Subjects: half-life (t½)
Pharmacokinetics (PK) Profile - MAD Clp | up to 28 days after last dose administration
  Pharmacokinetics Characteristics in Multiple Ascending Dose CF Subjects: plasma clearance (Clp)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan S Jafri, MD, FAAP, Study Director — Aridis Pharmaceuticals, Inc.; Alan H Cohen, MD, Study Director — Aridis Pharmaceuticals, Inc.
Locations (25):
- United States (25):
  - Research Site, Tucson, Arizona
  - Research Site, Long Beach, California
  - Research Site, Denver, Colorado
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
The Sponsor has not assessed whether to make individual participant data (IPD) available to other researchers.